CLINICAL TRIAL: NCT04027543
Title: Clinical Evidence for Association of Neoadjuvant Chemotherapy or Chemoradiotherapy With Efficacy and Safety in Patients With Resectable Esophageal Carcinoma (NewEC Study)
Brief Title: Neoadjuvant Chemotherapy or Chemoradiotherapy in Resectable Oesophageal Carcinoma（NewEC Study）
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-KS-2019-068
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Radiotherapy Side Effect; Chemotherapy Effect; Oesophageal Carcinoma; Effect of Drugs; Safety Issues
Keywords: Neoadjuvant chemoradiotherapy; Neoadjuvant chemotherapy; Resectable oesophageal carcinoma; Effective; Safety
MeSH Terms: conditions — Radiation Injuries; Esophageal Neoplasms | interventions — Neoadjuvant Therapy; Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Neoadjuvant chemoradiotherapy: Patients who had chemoradiotherapy before surgery.
  Interventions: Combination Product: Neoadjuvant chemoradiotherapy
- Neoadjuvant chemotherapy: Patients who had chemotherapy before surgery.
  Interventions: Drug: Neoadjuvant chemotherapy
- Surgery alone: Patients who only had oesophagectomy. Various surgical oesophagectomy methods were used, such as Ivor Lewis, transthoracic, three-hole, transhiatal, and left transthoracic. The appropriate surgical approach for each patient was chosen according to the tumour location, size, and depth.
  Interventions: Procedure: Oesophagectomy

INTERVENTIONS:
Combination Product: Neoadjuvant chemoradiotherapy — In most patients, the chemotherapy regimens before surgery were consisted of cisplatin combined with either fluorouracil or taxanes.
  Groups: Neoadjuvant chemoradiotherapy
Procedure: Oesophagectomy — Various surgical oesophagectomy methods were used, such as Ivor Lewis, transthoracic, three-hole, transhiatal, and left transthoracic,and the appropriate surgical approach for each patient was chosen according to the tumour location, size, and depth.
  Groups: Surgery alone
Drug: Neoadjuvant chemotherapy — In most patients, the chemotherapy regimens before surgery were consisted of cisplatin combined with either fluorouracil or taxanes.
  Groups: Neoadjuvant chemotherapy

SUMMARY:
To provide comprehensive efficacy and safety profiles of neoadjuvant chemoradiotherapy (NCRT) versus neoadjuvant chemotherapy (NCT) versus surgery alone in resectable oesophageal carcinoma.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy (NCT) or neoadjuvant chemoradiotherapy (NCRT) has been shown to be better than surgery alone in patients with resectable oesophageal carcinoma, but higher quality evidence is needed as new findings have emerged regarding this issue.Previous evidence-based findings and the current guidelines have not established a survival advantage of NCRT over NCT or an acceptable safety profile of the addition of radiotherapy to NCT; whether NCRT or NCT is more effective for the treatment of adenocarcinoma or squamous cell carcinoma of the oesophagus is unclear.This study aims to provide comprehensive efficacy and safety profiles of NCRT versus NCT versus surgery alone in resectable oesophageal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented untreated SCC or adenocarcinoma of the oesophagus or gastro-oesophageal junction.
* Patients clinically staged as stage I-III (T1-3, N0-1 and M0) as assessed by a contrast-enhanced multislice computed tomography (CT) scan, positron emission tomography, or endoscopic ultrasonography.
* Patients had an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

Exclusion Criteria:

* Patients had received any previous treatment for oesophageal cancer.
* Patients who were unsuitable for surgery because of comorbidities.
* Patients had evidence of distant metastatic disease by history and physical examination.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically documented untreated SCC or adenocarcinoma of the oesophagus or gastro-oesophageal junction that was clinically staged as stage I-III (T1-3, N0-1 and M0) as assessed by a contrast-enhanced multislice computed tomography (CT) scan, positron emission tomography, or endoscopic ultrasonography were eligible.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
  The OS was calculated as the time from the date of the histologically documented diagnosis to the date of death or the final follow-up.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  DFS was calculated from the date of R0 resection to the date of disease recurrence or death from any cause
R0 resection rate | Baseline
  R0 resection was defined as gross disease removed with negative margins (tumour-free resection margin).
Pathologic complete response (pCR) | Baseline
  pCR was defined as no evidence of residual tumour cells in the primary site and resected lymph nodes of the operative specimens.
30-day postoperative or in-hospital mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Herui Yao, PhD, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Haiyu Zhou, PhD, Principal Investigator — Guangdong Provincial People's Hospital; Michael Lanuti, PhD, Principal Investigator — Massachusetts General Hospital of Harvard Medical School
Locations (3):
- Massachusetts General Hospital of Harvard Medical School, Boston, Massachusetts, United States
- China (2):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No
The datasets used or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Zhou HY, Zheng SP, Li AL, Gao QL, Ou QY, Chen YJ, Wu ST, Lin DG, Liu SB, Huang LY, Li FS, Zhu HY, Qiao GB, Lanuti M, Yao HR, Yu YF. Clinical evidence for association of neoadjuvant chemotherapy or chemoradiotherapy with efficacy and safety in patients with resectable esophageal carcinoma (NewEC study). EClinicalMedicine. 2020 Jun 27;24:100422. doi: 10.1016/j.eclinm.2020.100422. eCollection 2020 Jul. PMID 32637899